CLINICAL TRIAL: NCT03781492
Title: Prospective REgistry of Stable Angina manaGEment and Treatment
Brief Title: Stable Angina Management and Treatment
Acronym: PRESAGE
Status: Recruiting | Type: Observational
Sponsor: Silesian Centre for Heart Diseases (Other)
Responsible Party: Principal Investigator, Mariusz Gasior, Clinical Professor, Silesian Centre for Heart Diseases
Other Study IDs: PRESAGE Registry
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Stable Angina; Coronary Artery Disease
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Prospective REgistry of Stable Angina manaGEment and Treatment (PRESAGE) is an observational study on an all-comer stable angina population hospitalised in a highly specialized cardiovascular centre with cardiac surgery facilities. The aim of the study is to assess the clinical characteristics, treatment modalities, early and long-term outcomes in this population.

DETAILED DESCRIPTION:
The Prospective REgistry of Stable Angina manaGEment and Treatment (PRESAGE) is a single-center, observational study recruiting consecutive patients with stable angina, who were diagnosed and treated in the 3rd Chair and Department of Cardiology in the Silesian Centre for Heart Diseases in Zabrze, Poland. The Silesian Centre for Heart Diseases is a highly specialised cardiology centre with cardiac surgery facilities

The main objective of the PRESAGE Registry is to clarify the overall clinical characteristics of patients with stable angina, their demographics and clinical profile, current management, early and long-term outcomes, with regard to the administered treatment.

The diagnosis of stable angina was based on clinical characterization, coronary angiography, and the current guidelines of the European Society of Cardiology. Patients with vasospastic and/or microvascular angina were also included to the registry. Performance of coronary angiography is the criterion of the enrolment in the registry.

Patients with acute coronary syndromes are excluded from the analysis.

Data collection is patient-based (not event-based).

Complete patient demographics: medical history, complete hospitalization data (diagnostic and therapeutic) and in-hospital results are collected in an electronic form by the attending physician. The patients are under constant follow-up for all-cause mortality and major cardiac adverse events.

ELIGIBILITY:
Inclusion Criteria:

* symptom based diagnosis of stable angina

Exclusion Criteria:

* acute coronary syndrome on admission
* ≤ 18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population is formed by all-comer patients hospitalized in cardiology ward with a diagnosis of stable angina.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2006-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with reported deaths from any cause | From date of inclusion until the date of death from any cause, assessed up to 5 year

SECONDARY OUTCOMES:
Number of participants with reported myocardial infarction | From date of inclusion until the date of first event, assessed up to 5 year
Number of participants with reported cerebrovascular insult | From date of inclusion until the date of first event, assessed up to 5 year
Number of participants with reported acute coronary syndrome driven revascularisation | From date of inclusion until the date of first event, assessed up to 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- 3rd Chair and Department of Cardiology of Silesian Centre for Heart Diseases, Zabrze, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No